CLINICAL TRIAL: NCT06040333
Title: The Effect of Dynamic Neuromuscular Stabilization Training in Dysfunctional Voiding : A Randomized Clinical Trial
Brief Title: Dynamic Neuromuscular Stabilization Training in Dysfunctional Voiding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Duygu Şahin Altaç, Principal investigator, MSc, PT, Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ssaka8
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Dysfunctional Voiding
Keywords: dysfunctional voiding; dynamic neuromuscular stabilization exercise
MeSH Terms: interventions — Exercise; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Neuromuscular Stabilisation Exercise (Experimental): The participants performed DNS exercises addition to standard therapy
  Interventions: Other: Exercise; Other: Standard therapy
- Standard therapy (Other): Patient education, massage, diaphragmatic breathing, kegel exercise
  Interventions: Other: Standard therapy

INTERVENTIONS:
Other: Exercise — Dynamic Neuromuscular Stabilisation Exercise
  Arms: Dynamic Neuromuscular Stabilisation Exercise
Other: Standard therapy — Patient education, massage, diaphragmatic breathing, kegel exercise

SUMMARY:
In this study, the effect of dynamic neuromuscular stabilization (DNS) exercise on urinary flow and quality of life in individuals with dysfunctional voiding was investigated. The 34 participants included in the study were randomized into two groups: the experiment in which DNS exercises were applied and the standard therapy group in which the manual application was applied. Uroflowmetry, Voiding Symptom Score (DVSS), Short Form-36 Quality of Life Assessment Short Form were applied to all participants at baseline and at week 6.

DETAILED DESCRIPTION:
In this study, the effect of dynamic neuromuscular stabilization (DNS) exercise on urinary flow and quality of life in individuals with dysfunctional voiding was investigated. This experimental study was conducted with patients who applied to UroKlinik in Istanbul between March 2021 and June 2023 and were diagnosed with dysfunctional voiding. The 34 participants included in the study were randomized into two groups: the experiment in which DNS exercises were applied and the standard therapy group in which the manual application was applied. Voiding Symptom Score (DVSS), Short Form-36 Quality of Life Assessment Short Form and Uroflowmetry test were applied to all participants before and at week 6.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with dysfunctional voiding,
* Being between the ages of 18-75,
* Not having a neurogenic bladder
* Not having a urinary tract infection
* Not having an obstacle to exercise,
* Accepting and signing the Approval Form,
* Not having undergone surgery in the last 6 months,

Exclusion Criteria:

* Not being cooperative
* Not being able to participate in the treatment,
* The use of drugs that will affect urination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Uroflowmetry - Maximum flow rate (Qmax) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *Qmax (mL/s): Qmax is the fastest stream measured in mL/s.
Uroflowmetry - Average flow rate (Qave) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *Qave (mL/s): Qave is the average stream measured in mL/s.
Uroflowmetry - Corrected maximum flow rate (cQmax) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *cQmax (mL/s/√ mL): cQmax is the precise assessment of fastest stream, especially at high volumes. Is it estimated Qmax/√ VV.
Uroflowmetry - Flow time (FT) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *FT (s): FT is the time over which measurable flow actually occurs.
Uroflowmetry - Voiding volume (VV) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *VV (ml): VV indicates the amount of voiding.
Uroflowmetry - Residual urine (RU) | at the baseline and at week 6.
  Uroflowmetry gives information about urine flow rate and voiding pattern.
  *RU (ml): RU is the amount of urine that is left behind in the bladder after you are done urinating.
Dysfunctional Voiding and Incontinence Symptom Score | at the baseline and at week 6.
  It gives information about voiding and incontinence symptoms. The questionnaire contains fourteen questions about symptoms and quality of life. The total score ranges from 0 to 35 and a score above 8.5 indicates abnormalities.
Short Form 36 | at the baseline and at week 6.
  It gives information about health related quality of life. The total score of the scale ranges from 0 to 100, and a high score indicates a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PhD, Study Director — Haliç University
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akbal C, Genc Y, Burgu B, Ozden E, Tekgul S. Dysfunctional voiding and incontinence scoring system: quantitative evaluation of incontinence symptoms in pediatric population. J Urol. 2005 Mar;173(3):969-73. doi: 10.1097/01.ju.0000152183.91888.f6. PMID 15711352
- [Result] Altunkol A, Abat D, Sener NC, Gulum M, Ciftci H, Savas M, Yeni E. Is urotherapy alone as effective as a combination of urotherapy and biofeedback in children with dysfunctional voiding? Int Braz J Urol. 2018 Sep-Oct;44(5):987-995. doi: 10.1590/S1677-5538.IBJU.2018.0194. PMID 30130020
- [Result] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695
- [Result] Haylen BT, Ashby D, Sutherst JR, Frazer MI, West CR. Maximum and average urine flow rates in normal male and female populations--the Liverpool nomograms. Br J Urol. 1989 Jul;64(1):30-8. doi: 10.1111/j.1464-410x.1989.tb05518.x. PMID 2765766
- [Result] Mahdieh L, Zolaktaf V, Karimi MT. Effects of dynamic neuromuscular stabilization (DNS) training on functional movements. Hum Mov Sci. 2020 Apr;70:102568. doi: 10.1016/j.humov.2019.102568. Epub 2020 Jan 13. PMID 31950895
- [Result] Zivkovic V, Lazovic M, Vlajkovic M, Slavkovic A, Dimitrijevic L, Stankovic I, Vacic N. Diaphragmatic breathing exercises and pelvic floor retraining in children with dysfunctional voiding. Eur J Phys Rehabil Med. 2012 Sep;48(3):413-21. Epub 2012 Jun 5. PMID 22669134